CLINICAL TRIAL: NCT05205564
Title: The Correlation of Stress and Coping, Resilience, and Compassion Fatigue of Nurses Staying on Front-line During COVID-19 Outbreak in Taiwan
Brief Title: Stress and Coping, Resilience, and Compassion Fatigue of Front-line Nurses During COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Piao-Yi Chiou, Associate Professor, National Taiwan University
Other Study IDs: 202106153RINB
Record Dates: First submitted 2022-01-21; First posted 2022-01-25 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: COVID-19 Pandemic; Stressor, Psychological; Mental Health Issue
Keywords: COVID-19; Front-line Nurses; Compassion Fatigue; Burnout; Stress Coping; Resilience
MeSH Terms: conditions — COVID-19; Stress, Psychological; Compassion Fatigue; Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is a cross-sectional research design. — No intervention will be involved in the study.

SUMMARY:
This is a cross-sectional research. The investigators plan to recruit about 250 front-line nurses who provided direct care to COVID-19 confirmed cases in a medical center in Taiwan. Online querstionnaires are used to collect the data. The relationship between variables such as stressors related to COVID-19, coping status, resilience, and compassion fatigue of participants will be analysis to provide the direction of nurses' mental health-related interventions.

DETAILED DESCRIPTION:
This project aims to identify the prevalence of compassion fatigue and the coping strategies for the nurses who work on the frontline of healthcare and are responsible for caring for patients with COVID-19 in Taiwan. The investigators planed to carry a cross-sectional study by a reliable and valid online questionnaire to explore the stressors related to COVID-19, coping status, resilience, and compassion fatigue of nurses who had the experience of caring for the COVID-19 confirmed cases in a medical center during the community outbreak in Taiwan from May 2021. Online questionnaires are used to collect the data. About two hundred and fifty nurses will be recruited, and the data will be analyzed by descriptive statistics, correlation statistics and Hayes's PROCESS model 6. It is expected that the research results can understand the current status and relationship of compassion fatigue, resilience and the adaptability of clinical nurses who are caring for the COVID-19 confirmed cases. The results can be contributed to develop the direction of nurses' mental health-related interventions during pandemic of emerging contagious disease.

ELIGIBILITY:
Inclusion Criteria:

* Above/include 20-year-old.
* Those who can operate mobile communication software or computers and can fill in online questionnaires.
* Clinical nurses who had provided nursing care for COVID-19 confirmed cases from May 2021.

Exclusion Criteria:

* Those who did not provide nursing care for COVID-19 confirmed cases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinical nurses who have been or are still working in hospital, and have directly cared for COVID-19 confirmed cases from May 2021.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Interaction effect between research variables | six months to collect and analysis data.
  Factors including "stressors related to COVID-19", "stress coping", "resilience", and "compassion fatigue" have interaction effect.
Moderation effect between research variables | six months to collect and analysis data.
  Both "stress coping" and "resilience" moderate the strength relationship between "stressors" and "compassion fatigue".

CONTACTS AND LOCATIONS:
Overall Officials: YI-CHEN YEH, Bachelor, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei, Zhongzheng Dist.
  - School of Nursing of National Taiwan University, Taipei